CLINICAL TRIAL: NCT03963167
Title: The Impact on the Health Status and Adherence in a Real-life Setting of Italian Patients With Chronic Obstructive Pulmonary Disease in Treatment With Trimbow® pMDI b.i.d.: a 12-month Prospective Observational Study
Brief Title: Triple Therapy in Real-life: Impact on Adherence and Health Status (TRITRIAL)
Status: Completed | Type: Observational
Sponsor: Chiesi Italia (Industry)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Other Study IDs: DFIDM-1802
Record Dates: First submitted 2019-05-14; First posted 2019-05-24 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: COPD
Keywords: COPD; Adherence; HRQoL determinants
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient in treatment with BDP/FF/G fixed combination
  Interventions: Drug: BDP/FF/G fixed combination

INTERVENTIONS:
Drug: BDP/FF/G fixed combination — Fixed combination of Inhaled Corticosteroid (ICS) / Long-acting β2-agonist (LABA) / long-acting muscarinic antagonist (LAMA) that contains Beclometasone dipropionate (BDP), Formoterol fumarate (FF) and Glycopyrronium (G).
  Other Names: Trimbow

SUMMARY:
The mean objectives are to evaluate the impact of BDP/FF/G fixed combination on health-status and adherence

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study;
2. Adult patients of either sex aged ≥ 40 years;
3. Patients with diagnosis of moderate to very severe COPD according to Gold Initiative for Chronic Obstructive Lung Disease (GOLD) updated 2019 (GOLD Stage 2-4);
4. COPD assessment test (CAT) score ≥ 10 at initiation of BDP/FF/G fixed combination;
5. History of >1 moderate or severe COPD exacerbation during the previous year.
6. Patients in treatment with BDP/FF/G as per local clinical practice and according to Trimbow® Summary of Product Characteristics (SmPC).

Exclusion Criteria:

1. According on Investigator's judgement, patients unable to comply with the requirements of the study (e.g. inability to attend all the planned study visits according to the time limits included) or patients with poorly controlled concomitant severe diseases or conditions that could interfere with the study participation;
2. Participation in an interventional clinical trial within 30 days prior to enrolment into the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients with symptoms and history of exacerbations despite of maintenance therapy
Sampling Method: Non-Probability Sample
Enrollment: 661 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Change in COPD Assessment Test (CAT) score | 12 months
  CAT consists of 8 items scored on a scale of 1 to 5, with a total score range of 0-40. A higher score denotes a more severe impact of COPD on the patient's life.

SECONDARY OUTCOMES:
Change in COPD Assessment Test (CAT) score | 6 months
  CAT consists of 8 items scored on a scale of 1 to 5, with a total score range of 0-40. A higher score denotes a more severe impact of COPD on the patient's life.
Change in 12-item Test of Adherence to Inhalers (TAI-12) score | 6 and 12 months
  TAI comprises a patient domain (including 10 items) and a healthcare professional domain (including 2 items). Each item ranges from 1 (lowest adherence) to 5 (highest adherence) points. The patient domain score ranges from 10 to 50. Adherence is rated as good (score =50), intermediate (score = 46-49), or poor (score ≤45). The questions for healthcare professionals are scored with 1 or 2 points (poor or good knowledge of the regimen and/or inhalation technique).
Change in COPD and Asthma Sleep Impact Scale (CASIS) score | 6 and 12 months
  It is a self-administered 7-item scale scored on a five-point scale ranging from 0 if the item never applies, to 4 if the item applies very often. A total raw score is produced from the sum of the seven individual scores which is then linearly transformed to a 0-100 total scale score. Higher scores representing greater sleep deterioration in the previous week.
Change in EuroQoL score | 6 and 12 months
  Il consists of 2 pages, a descriptive system and a visual Analogue scale. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each dimension having 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.The VAS records the respondent's self-rated health on a 10 cm vertical VAS with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
Change of an 8-item questionnaire on satisfaction and usability of the device score from baseline (Visit 1) | 6 and 12 months
  it contains 8 questions, each scored on a 0-5 Likert scale, which range from 0 (fully disagree) to 5 (fully agree), for a total maximum score of 40. Higher scores indicate a higher ease of use and satisfaction with the inhaler
Forced Expiratory Volume in the first second (FEV1, L) | Baseline, 6 and 12 months
Forced Vital Capacity (FVC, L) | Baseline, 6 and 12 months
Mean forced expiratory flow between 25% and 75% of the FVC (FEF25-75) | Baseline, 6 and 12 months
  Taken from the test with the highest values of FEV1 and FVC
Ratio FEV1/FVC | Baseline, 6 and 12 months
  Derived from these highest values of each parameter
Use of rescue medication | Baseline, 6 and 12 months
  Use of rescue medication
Exacerbations | Baseline, 6 and 12 months
  Moderate to severe exacerbations
Adverse events | Baseline, 6 and 12 months
  Number of adverse events
Economic resources consumption | Baseline, 6 and 12 months
  Number of hospitalizations, ER access, unscheduled visits

CONTACTS AND LOCATIONS:
Overall Officials: Luca Richeldi, MD, Principal Investigator — Policlinico Gemelli, Roma (Italy)
Locations (1):
- Fondazione Policlinico Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No